CLINICAL TRIAL: NCT05436574
Title: Impact of the Implementation of Dance Therapy Workshops on the Quality of Life of Dependent Elderly People Institutionalized Within the Establishments of the Univi Group: Longitudinal Intervention Study
Brief Title: Impact of the Implementation of Dance Therapy Workshops on the Quality of Life of Dependent Elderly People Institutionalized Within the Establishments of the Univi Group
Acronym: Unidance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Médical Porte Verte (Other)
Responsible Party: Principal Investigator, Valérie BRENIERE, Study coordinator, Centre Médical Porte Verte
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A01255-38
Record Dates: First submitted 2022-06-17; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Dance Therapy Workshop
MeSH Terms: interventions — Dance Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before/after study (Other): Before/after study to measure the effects of the implementation of a dance therapy activity on the quality of life of the elderly population
  Interventions: Other: Dance therapy

INTERVENTIONS:
Other: Dance therapy — Before/after study to measure the effects of the dance therapy activity on the quality of life of the elderly population housed in the establishments of UNIVI group.

SUMMARY:
Dance is a multimodal activity involving motor, cognitive, sensory and sensory-motor skills as well as emotional and social skills. A growing body of research shows that the creative arts and physical exercise are able to alleviate disability, improve social interactions, and slow the progression of Alzheimer's disease and related disorders.

The Associative Group UNIVI wants to evaluate through this study the effects of the practice of dance on the quality of life of the people accommodated in its USLD and EHPAD

DETAILED DESCRIPTION:
This research is an interventional study involving the human person of category 2 involving only minimal risks and constraints, it is multicentric and longitudinal prospective. This is a before/after study to measure the effects of the implementation of a dance therapy activity on the quality of life of the elderly population housed in the 30 establishments of the univi group.

The dance therapy will be deployed in all the medico-social establishments participating in the study over a period of 12 weeks.

To do this, dance therapists will be recruited to provide these classes.

The dance-therapy will be carried out:

* in groups of 10 to 12 people who have given their informed consent,
* at least twice a week per group,
* over a period of 30 to 45 minutes maximum twice a week for 3 months. Several groups per establishment can be planned depending on the number of people who can and want to be included in the dance workshop.

  940 participant in the study will be inclued and followed at 1 month, 3 months and 6 months after the end of the dance therapy workshops.

ELIGIBILITY:
Inclusion Criteria:

* People aged over 60
* Dependent elderly people residing in EHPAD or USLD including people under guardianship and curatorship
* People having signed an informated and weitten consent
* People with a minimum of language skills to understand instructions and simple questions

Exclusion Criteria:

* Participants in palliative care
* Contraindication to the practice of dance
* Severe cognitive and/or behavioral disorders that do not allow you to follow a dance workshop
* Permanent bed rest
* Non-affiliation to a social security scheme

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
QOL-AD NH scale | Eight months
  The QOL-AD is a brief 13-item measure designed specifically to obtain an assessment of the patient's quality of life from both the patient and the caregiver.
  It was developed for people with dementia, based on feedback from patients, caregivers and experts, to maximize construct validity and ensure measurement focuses on areas of quality of considered important in older adults with cognitive impairment The measurement of 13 items, rated on a four-point scale, of which 1 is poor and 4 excellent. Total partitions range from 13 to 52.

SECONDARY OUTCOMES:
Tinetti test: assessement of walking and balance | Eight months
  The Tinetti test is an effective and reproductible tool for the assessement of the risk of falling, its administration time is approximately 5 to 10 minutes and evaluates static and dynamic balance
Get up and Go test | Eight months
  This test evaluates the transfers sitting, standing, walking and changes of direction of the person. . Interpretation: risk of falling if score greater than or equal to 9
Time up and Go test | Eignt months
  The time up and go test is the timed version of the get up and go test. The subject seated on a chair must get up, walk 3 meters in front of him, return to his chair and sit down. The score is given by the time in seconds.
  Interpretation: risk of falling if the score is greater than or equal to 21 seconds.
NPI-ES: NEUROPSYCHIATRIC INVENTORY | Eight months
  assesses the presence of behavioral problems in people with dementia. . a score of Ten behavioral domains and 2 neurovegetative variables are taken into account.
The mini GDS | Eight months
  The mini GDS (Geriatric Depression Scale) aims to identify the person's risk of depression. It consists of 4 simple questions that must be answered with "yes" or "no".